CLINICAL TRIAL: NCT03131791
Title: Radial Extracorporeal Shock Wave Versus Botulinum Toxin A in the Treatment of Post-Stroke Upper Limb Spasticity: A Randomized Non-Inferiority Trial
Brief Title: Comparing the Radial Extracorporeal Shock Waves and Botulinum Toxin Injection for Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Gwo-Chi Hu,PHD, PHD, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16MMHIS066e
Record Dates: First submitted 2017-04-21; First posted 2017-04-27 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Post-Stroke Upper Limb Spasticity
Keywords: Extracorporeal Shock Wave; Spasticity in stokes; Botulinum toxin
MeSH Terms: interventions — Extracorporeal Shockwave Therapy; Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: group A : shock wave, group B: Botulinum Toxin Injection
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- shock wave (Experimental): The interventions were focused in the hypertonic muscles of the upper limb of 3000 impulses, a pressure of 1.5 bar and frequency of 5Hz were used to treat the biceps brachii, flexor carpi ulnaris and flexor carpi radialis, mainly in the middle of the belly.
  Interventions: Device: Shock Wave
- Botulinum toxin A (Experimental): We performed BoNT-A 500 unit in 2cc 0.9% normal saline at biceps brachii, flexor carpi ulnaris and flexor carpi radialis, mainly in the middle of the belly.
  Interventions: Drug: Botulinum toxin A

INTERVENTIONS:
Device: Shock Wave — 42 chronic stroke patients with upper limb spasticity were randomly assigned to receive either 1 session of ESWT per week for 3 consecutive weeks or BoNT-A injection. The biceps, flexor carpi radialis, and flexor carpi ulnaris muscles were treated. Assessments were performed at baseline and at 1, 4, and 8 weeks after the intervention. The primary outcome measure was the change in the Modified Ashworth Scale (MAS) score for the elbow from the baseline to after 4 weeks of treatment.
  Arms: shock wave
Drug: Botulinum toxin A — 42 chronic stroke patients with upper limb spasticity were randomly assigned to receive either 1 session of ESWT per week for 3 consecutive weeks or BoNT-A injection. The biceps, flexor carpi radialis, and flexor carpi ulnaris muscles were treated. Assessments were performed at baseline and at 1, 4, and 8 weeks after the intervention. The primary outcome measure was the change in the Modified Ashworth Scale (MAS) score for the elbow from the baseline to after 4 weeks of treatment.
  Arms: Botulinum toxin A

SUMMARY:
Botulinum toxin type A (BoNT-A) is widely used in the clinics to reduce spasticity and improve upper limb function for post-stroke patients. However, there were no studies to compare the effect of rESWT and BoNT-A injection for treatment on spasticity.

DETAILED DESCRIPTION:
Botulinum toxin type A (BoNT-A) is widely used in the clinics to reduce spasticity and improve upper limb function for post-stroke patients. However, the treatments of BoNT-A injection are associated with high cost and invasive treatment. Recent studies have showed that radial extracorporeal shock wave (rESWT) is a novel, effective and safety treatment method for the spasticity. However, there were no studies to compare the effect of rESWT and BoNT-A injection for treatment on spasticity.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18-80 year-old
2. The onset of stroke must be at least 6 months previously
3. Spasticity measured as Modified Asthow Scale more(MAS) than 1+
4. Signed informed consent form

Exclusion Criteria:

1. Patients with marked contractures in the elbow and wrist (MAS>4)
2. Resistant hypertension, coagulation disorders, malignant tumors, pregnancy, pacemakers, cognitive disorders
3. Prior or planned treatment with phenol or alcohol nerve blocks, intrathecal baclofen, or BoNT-A injection within the six months preceding the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
The change of spasticity of elbow | Between baseline and 4 weeks post-treatment
  Modified Ashworth Scale (MAS) for spasticity

SECONDARY OUTCOMES:
The change of Tardieu scale scores for the elbow and wrist | Between baseline and 1, 4,8 weeks post-treatment
  Tardieu scale scores for spasticity
The change of upper limb function | Between baseline and 1,4,8 weeks post-treatment
  The Fugl-Meyer Assessment (FMA) for upper limb function

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Wu YT, Yu HK, Chen LR, Chang CN, Chen YM, Hu GC. Extracorporeal Shock Waves Versus Botulinum Toxin Type A in the Treatment of Poststroke Upper Limb Spasticity: A Randomized Noninferiority Trial. Arch Phys Med Rehabil. 2018 Nov;99(11):2143-2150. doi: 10.1016/j.apmr.2018.05.035. Epub 2018 Jul 4. PMID 30392753

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT03131791/Prot_SAP_000.pdf